CLINICAL TRIAL: NCT05035654
Title: BEACON: A Phase II, Patient-blinded, Two-part, Randomized, Parallel-group Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of LYR-220 in Chronic Rhinosinusitis (CRS) Patients Who Have Had a Prior Ethmoidectomy
Brief Title: LYR-220 for Adult Subjects With Chronic Rhinosinusitis (BEACON Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lyra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYR-220-2021-001
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Chronic Sinusitis; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1: Treatment Arm LYR-220 Design 1 (Experimental): Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 1
  Interventions: Drug: LYR-220 Design 1 (Part 1 only)
- Part 1 and Part 2: Treatment Arm LYR-220 Design 2 (Experimental): Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
  Interventions: Drug: LYR-220 Design 2 (Part 1 and Part 2)
- Part 2: Treatment Arm Bilateral sham procedure control (Sham Comparator): Bilateral sham procedure control
  Interventions: Drug: Bilateral sham procedure control (Part 2)

INTERVENTIONS:
Drug: LYR-220 Design 1 (Part 1 only) — LYR-220 drug matrix (mometasone furoate 7500 µg) Design 1
  Arms: Part 1: Treatment Arm LYR-220 Design 1
Drug: LYR-220 Design 2 (Part 1 and Part 2) — LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
  Arms: Part 1 and Part 2: Treatment Arm LYR-220 Design 2
Drug: Bilateral sham procedure control (Part 2) — Bilateral sham procedure control
  Arms: Part 2: Treatment Arm Bilateral sham procedure control

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics and efficacy of two LYR-220 designs in symptomatic adult chronic rhinosinusitis (CRS) subjects who have had a prior functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
This is a Phase II, Patient-blinded, Two-part, Randomized, Parallel-group Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of LYR-220. The study will consist of two parts: Part 1 will enroll up to 10 patients and is open label. Part 2 is randomized, sham controlled and will enroll approximately 40 patients. The study follow-up duration is 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis.
* Has had a prior bilateral total ethmoidectomy.
* Has computed tomography (CT) ethmoid cavity opacification.
* Has a Sinonasal Outcome Test (SNOT-22) ≥ 20 at Screening Visit.
* Minimum cardinal symptom score.
* Has been informed of the nature of the study and has provided written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site or regulatory authority if applicable by national law.
* Agrees to comply with all study requirements.

Exclusion Criteria:

* Pregnant or breast feeding.
* Known history of hypersensitivity or intolerance to corticosteroids.
* History or clinical evidence or suspicion of invasive fungal sinusitis, allergic fungal rhinosinusitis, or atrophic rhinitis.
* Known history of hypothalamic pituitary adrenal axial dysfunction.
* Had dental procedure/implant on maxillary dentition within 4 weeks of the Screening visit.
* Past or present functional vision in only one eye.
* Past, present, or planned organ transplant or chemotherapy with immunosuppression.
* With prior cataract surgery or presence (in either eye) of posterior subcapsular cataract of grade 2 or higher, nuclear cataract of grade 3 or higher, or cortical cataract of grade 2 or higher or involving a minimum of center optic zone of 3 mm diameter.
* Ethmoidectomy that was unilateral or partial.
* Currently participating in an investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (21):
  - Lyra Investigational Site, Carlsbad, California
  - Lyra Investigational Site, La Mesa, California
  - Lyra Investigational Site, Roseville, California
  - Lyra Investigational Site, Torrance, California
  - Lyra Investigational Site, Chicago, Illinois
  - Lyra Investigational Site, New Albany, Indiana
  - Lyra Investigational Site, Louisville, Kentucky
  - Lyra Investigational Site, Marrero, Louisiana
  - Lyra Investigational Site, Baltimore, Maryland
  - Lyra Investigational Site, New Hyde Park, New York
  - Lyra Investigational Site, New York, New York
  - Lyra Investigational Site, Chapel Hill, North Carolina
  - Lyra Investigational Site, Winston-Salem, North Carolina
  - Lyra Investigational Site, Bethlehem, Pennsylvania
  - Lyra Investigational Site, Orangeburg, South Carolina
  - Lyra Investigational Site, Spartanburg, South Carolina
  - Lyra Investigational Site, Fort Worth, Texas
  - Lyra Investigational Site, McKinney, Texas
  - Lyra Investigational Site, San Antonio, Texas
  - Lyra Investigational Site, South Ogden, Utah
  - Lyra Investigational Site, Spokane, Washington
- Australia (3):
  - Lyra Investigational Site, Bedford Park
  - Lyra Investigational Site, Brisbane
  - Lyra Investigational Site, Melbourne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 subjects were randomized but did not receive the investigational product and are not included in the total count
Groups:
- Part 1: LYR-220 Design 1: Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 1
  LYR-220 Design 1: LYR-220 drug matrix (mometasone furoate 7500 µg) Design 1
- Part 1 and Part 2: LYR-220 Design 2: Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
  LYR-220 Design 2: LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
- Part 2:Bilateral Sham Procedure: Bilateral sham procedure control
  Bilateral sham procedure control: Bilateral sham procedure control
Period: Overall Study
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2:Bilateral Sham Procedure
Started | 3 | 24 | 21
Completed | 2 | 22 | 17
Not Completed | 1 | 2 | 4
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Bilateral Dislodgement | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 2: Bilateral Sham Procedure: Bilateral sham procedure control Bilateral sham procedure control: Bilateral sham procedure control
- Total: Total of all reporting groups
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure | Total
Number analyzed (Participants) | 3 | 24 | 21 | 48
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 subjects were randomized but did not receive the investigational product.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 2 | 23 | 18 | 43
    >=65 years | 1 | 1 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (14.98) | 48 (12.91) | 55 (11.29) | 51 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 subjects were randomized but did not receive the investigational product.
  Participants
    Female | 1 | 16 | 11 | 28
    Male | 2 | 8 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 subjects were randomized but did not receive the investigational product
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 0 | 1 | 2 | 3
    White | 3 | 22 | 18 | 43
    More than one race | 0 | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 20 | 21 | 44
  Australia | 0 | 4 | 0 | 4
BMI [Mean (Standard Deviation); unit: kg/m²] — Population: Subjects with non-missing height and/or weight.
  kg/m²
    number analyzed (Participants) | 2 | 21 | 19 | 42
    (all) | 35.35 (6.69) | 30.65 (5.68) | 33.71 (8.63) | 32.26 (7.23)

OUTCOME MEASURES:

1. Primary Outcome: Product-related Unexpected Serious Adverse Events
Description: Product-related unexpected serious adverse events
Time Frame: Through Week 28
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
Number analyzed (Participants) | 3 | 24 | 21
Participants | 0 | 0 | 0

2. Primary Outcome: Plasma MF Concentrations
Description: Plasma MF concentrations at 1 hour post study treatment administration and at Days 2 or 3, days 5 or 8, and Weeks 4,12,16 or 20, 24 and 25.
  The PK analysis will be performed based on subjects with available plasma MF concentration data post Day 1 administration procedure.
Time Frame: Through Week 25
Population: PK Analysis Set Design 1- Part 1, PK Analysis Set Design 2 - Part 1; PK Analysis Set Design 2 - Part 2
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Part 1: Treatment Arm LYR-220 Design 1: Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 1
  LYR-220 Design 1: LYR-220 drug matrix (mometasone furoate 7500 µg) Design 1
- Part 1: Treatment Arm LYR-220 Design 2; Part 2: Treatment Arm LYR-220 Design 2: Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
  LYR-220 Design 2: LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
Arm/Group | Part 1: Treatment Arm LYR-220 Design 1 | Part 1: Treatment Arm LYR-220 Design 2 | Part 2: Treatment Arm LYR-220 Design 2
Number analyzed (Participants) | 3 | 3 | 21
pg/mL
  1-Hour Post: number analyzed (Participants) | 2 | 0 | 16
  1-Hour Post | 11.04 (0.04) |  | 18.11 (13.09)
  Day 2: number analyzed (Participants) | 2 | 1 | 15
  Day 2 | 40.86 (5.98) | 135.83 | 61.02 (23.98)
  Day 3: number analyzed (Participants) | 1 | 2 | 5
  Day 3 | 97.77 | 55.86 (28.70) | 46.00 (26.05)
  Day 5: number analyzed (Participants) | 0 | 0 | 6
  Day 5 |  |  | 44.16 (19.60)
  Day 8: number analyzed (Participants) | 2 | 3 | 14
  Day 8 | 68.34 (38.67) | 72.31 (19.15) | 58.87 (21.36)
  Week 4: number analyzed (Participants) | 3 | 3 | 19
  Week 4 | 40.41 (25.99) | 68.90 (5.19) | 61.31 (34.97)
  Week 12: number analyzed (Participants) | 3 | 3 | 19
  Week 12 | 15.14 (4.26) | 68.00 (20.96) | 50.17 (17.79)
  Week 16: number analyzed (Participants) | 0 | 1 | 9
  Week 16 |  | 70.940 | 31.26 (17.06)
  Week 20: number analyzed (Participants) | 2 | 2 | 9
  Week 20 | 7.58 (5.31) | 22.6 (1) | 20.17 (8.49)
  Week 24: number analyzed (Participants) | 2 | 3 | 18
  Week 24 | 2.08 (2.14) | 11.52 (8.77) | 11.18 (12.96)
  Week 25: number analyzed (Participants) | 0 | 0 | 2
  Week 25 |  |  | NA (NA) — Statistics at any individual timepoint were calculated if at least half of the subjects have valid values (ie not missing, quantifialble and not outside collection window). Actual sampling times that were outside the sampling time windows were excluded from concentration summary.

3. Secondary Outcome: Adverse Events
Description: Percentage of subjects reporting treatment-emergent adverse events
Time Frame: Through Week 28
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
Number analyzed (Participants) | 3 | 24 | 21
Participants | 1 | 23 | 16

4. Secondary Outcome: Endoscopic Findings
Description: Percentage of subjects with newly identified or worsened endoscopic findings in the ethmoid cavity (mild, moderate, or severe)
Time Frame: Through Week 25
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
Number analyzed (Participants) | 3 | 24 | 21
Participants | 0 | 6 | 3

5. Secondary Outcome: Ophthalmic Assessment: Intraocular Pressure (IOP)
Description: Percentage of subjects with clinically significant increase in IOP
Time Frame: Through Week 25
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
Number analyzed (Participants) | 3 | 24 | 21
participants
  IOP in 1 or both eyes >23 mm Hg at Post Baseline | 0 | 0 | 0
  An increase of IOP from Baseline in 1 or both eyes >=10 mm Hg | 0 | 0 | 0

6. Secondary Outcome: Ophthalmic Assessment: Cataract
Description: Percentage of subjects with newly identified or worsened cataract in one or both eyes
Time Frame: Through Week 25
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
Number analyzed (Participants) | 3 | 24 | 21
Participants
  Newly Identified Cataract | 0 | 1 | 0
  Worsened Cataract | 0 | 1 | 0

7. Secondary Outcome: Improving Chronic Rhinosinusitis (CRS) Specific Quality of Life as Per the 22-item Sino-nasal Outcome Test (SNOT-22) Questionnaire
Description: The 22-item Sino-Nasal Outcome Test (SNOT-22) questionnaire is a 22-item disease-specific quality of life instrument validated for use in CRS. Each symptom is scored as it has been over the past 2 weeks on a 6-point scale as follows: 0 = no problem, 1 = very mild problem, 2 = mild or slight problem, 3 = moderate problem, 4 = severe problem, 5 = problem as bad as it can be.
  The outcome measure is change from baseline in total patient-reported outcome score. The SNOT-22 total score is the sum of individual scores and ranges from 0 to 110. Higher scores indicate higher severity of symptoms.
Time Frame: Through Week 28
Population: Efficacy Analysis Set - Part 2
Measure: Mean (Full Range); unit: Change from Baseline in SNOT-22 score
Groups:
- Part 2 LYR-220 Design 2: Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2 LYR-220 Design 2: LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
- Part 2 Bilateral Sham Procedure: Bilateral sham procedure control Bilateral sham procedure control: Bilateral sham procedure control
Arm/Group | Part 2 LYR-220 Design 2 | Part 2 Bilateral Sham Procedure
Number analyzed (Participants) | 13 | 9
Change from Baseline in SNOT-22 score | -30.1 [-74 to -2] | -4.0 [-34 to 32]

8. Secondary Outcome: Change From Baseline in the Average Composite Score Over the Preceeding 7 Days of the 3 Cardinal Symptoms (3CS)
Description: Change from baseline in the average composite score over the preceeding 7 days of the 3 Cardinal Symptoms (3CS).The 3CS include: nasal blockage/obstruction/congestion, facial pain/ pressure, and anterior/posterior nasal discharge. The diary is completed daily by study participants throughout the study. Each symptom/each question is scored daily on a 0-3 scale as follows: 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The 3CS total score ranges from 0-9, with higher scores indicating worse symptoms.
Time Frame: Through Week 28
Population: Efficacy Analysis Set - Part 2
Measure: Mean (Standard Deviation); unit: Change from Baseline in 3CS Score
Groups:
- Part 2: LYR-220 Design 2: Bilateral insertion of LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2 LYR-220 Design 2: LYR-220 drug matrix (mometasone furoate 7500 µg) Design 2
Arm/Group | Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
Number analyzed (Participants) | 21 | 21
Change from Baseline in 3CS Score | -1.68 (2.33) | -0.48 (2.1)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported from Day 1 through Week 28 (~ 7 months).
Description: Standard definition of adverse events and serious adverse events was used in the trial.
  All events were assesed for relationship to the study product and study procedure.
Arm/Group | Part 1: LYR-220 Design 1 | Part 1 and Part 2: LYR-220 Design 2 | Part 2: Bilateral Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 1/3 | 21/24 | 9/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: LYR-220 Design 1 (N=3) | Part 1 and Part 2: LYR-220 Design 2 (N=24) | Part 2: Bilateral Sham Procedure (N=21)
Sinusitis (Infections and infestations) | 0 (0) | 8 (11) | 4 (4)
Acute Sinusitis (Infections and infestations) | 1 (1) | 6 (9) | 2 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Nasal Odour (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except as approved by Sponsor, single center data will not be published before multicenter data, unless >1 year has elapsed since completion of the Study. PI may publish single center data provided that PI shall: i) provide a copy of the publication to Sponsor at least 60 days in advance of submission for publication; ii) delete Sponsor Confidential Information and make other reasonable changes; and iii) delay submission by up to 90 additional days to permit intellectual property filings.

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT05035654/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT05035654/SAP_001.pdf